CLINICAL TRIAL: NCT00805662
Title: Nasal Oxcytocin Fails to Increase Pregnancy Rate of IUI
Brief Title: Nasal Oxcytocin During IUI
Acronym: Oxy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Organon GmbH (former name) (Unknown); Essex Pharma GmbH (Industry)
Responsible Party: Prof. Dr. Klaus Friese, Department of Obstetrics and Gynecology, Campus Grosshadern, LMU
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 355/02
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Idiopathic Infertility
Keywords: IUI; oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxytocin (Experimental): Intranasal oxytocin during IUI
  Interventions: Drug: oxytocin, placebo

INTERVENTIONS:
Drug: oxytocin, placebo — intranasal oxytocin during intrauterine insemination
  Other Names: Synthocinon

SUMMARY:
Placebo-controlled study. Application of nasal oxytocin (8 IU) during intrauterine insemination in 86 patients.

DETAILED DESCRIPTION:
Between 2004 and 2007, 86 patients with primary or secondary infertility were enrolled in this prospective, randomized, double-blinded study in our tertiary-care infertility center. A total of 132 homologous intrauterine insemination (IUI) cycles (mean: 1.5 cycles) was performed. All patients gave informed consent. The study was approved by the Human Ethics Committee of the Medical Faculty of the Ludwig-Maximilians-University (LMU) Munich and the German Federal Institute for Drugs and Medical Products (BfArM) (Bundesinstitut für Arzneimittel und Medizinprodukte) consented to the study.

Inclusion criteria for couples were idiopathic infertility, polycystic ovary syndrome (PCOS) and / or male subfertility (table 1). Maximum female age was 42 years. Infertility workup included a standard gynecological examination with a transvaginal sonography using a 7.5 MHz probe. Patients displaying signs or symptoms of anomalies such as uterine fusion defects, submucosal fibroids, active endometriosis or acute inflammation were excluded from the study. Further prerequisites were endocrine serum parameters (FSH, LH, estradiol, testosterone, SHBG, DHEA-S, Prolaktin, TSH) from cycle day 2-5 within the normogonadotropic range with no evidence of hyperandrogenemia, thyroid dysfunction or hyperprolactinemia. 15 patients were diagnosed with polycystic ovary syndrome (PCOS) according to the Rotterdam ESHRE/ASRM Consensus Workshop Group (26). In all patients fallopian tubes were documented to be patent by sonographic contrast hysterosalpingography (Echovist® 200, Bayer Vital GmbH, Leverkusen, Germany) or by chromo-laparoscopy. Infections with Hepatitis B and C and HIV were excluded in all couples by negative serological tests. In all patients protective titers against rubella virus were confirmed.

IUI was performed in natural (n=31, 23%) or stimulated cycles (n=101, 77%). Stimulation was done with daily s.c. 37 IU or 50 IU of recombinant FSH (Puregon, Organon GmbH, Oberschleißheim, Germany) starting on day 3 to day 5 of the menstrual cycle. Cycles were monitored by repeated transvaginal sonography and determination of serum estradiol and LH. Ovulation induction (OI) was done by 5.000 IU hCG (Predalon, Organon GmbH, Oberschleißheim, Germany) s.c. or 250 μg recombinant hCG (Ovitrelle, Serono GmbH, Unterschleißheim, Germany) s.c. as soon as one of maximum three follicles reached a mean diameter of 20 mm or LH exceeded 10 mIU/mL in combination with a follicle mean diameter of at least 16 mm. IUI was done 24h-36h after OI. Data on uterine, ovarian and endocrine parameters at the time of ovulation induction (OI) are summarized in table 2.

Homologous semen samples were gained by masturbation after an abstinence time of 3-5 days. After liquification for 30 min analysis of semen parameters were carried out according to the World Health Organization guidelines (27). Details on results are summarized in table 2. Sperm morphology was analysed according to WHO guidelines in at least one semen analysis preceding this study not more than 3 months. The sperm preparation was conducted utilizing density gradient separation as described in the WHO manual (27). Sil Select (FertiPro N.V., Beernem, Belgium) was used instead of Percoll as recommended in the WHO manual (27). The density gradient (90%/45%) achieved separation of sperm after centrifugation at 500 g for 20 minutes. The pellet was washed in 5.0 mL Universal IVF Medium (Medi Cult, Jyllinge, Denmark), centrifuged for 5 minutes at 500 g and resuspended in a total volume of 0.3 mL. After processing, semen was evaluated for sperm concentration and motility. Only couples with a total progressive motile sperm count (TPMC) of at least 1 million in the processed sperm suspension were included in the study. Data are summarized in table 2.

Oxytocin and placebo, filled in identical nasal spray applicators labelled with "A" or "B", were delivered by the pharmacy department of LMU-Klinikum, Campus Grosshadern. Probes were blinded to the clinical staff and the patients. The verum consisted of Synthocinon®-Spray (Novartis Pharma GmbH, Nürnberg, Germany). According to the manufacturer one nasal spray pump consists of 4 IU of oxytocin. In addition the verum contained chlorobutanol, methyl-4-hydroxybenzoat and propyl-4-hydroxybenzoat for preservation. Placebo consisted of isotonic NaCl solution with 0.01 % benzalkoniumchloride und 0.1% Na-EDTA for preservation. The nasal sprays were kept at 4°C and replaced monthly. Patients were randomly assigned to either group A or group B (double-blinded) by using a computer generated randomization list. Codes for A and B were broken after the last study patient had completed the pregnancy test. Data on patient variables in both groups are summarized in table 2. All patients were asked to squeeze the spray into the air for control of the pump mechanism and then to apply two snuffs (=8 IU oxytocin) of nasal spray labelled with A and B respectively into one nostril directly after IUI.

Ten minutes after completion of the IUI patients were asked to fill out a form documenting possible side effects. Each of the following complaints was asked to be quantified in a scale from level 1 (=no side effect) to level 10 (=maximum side effect): lower abdominal pain, nasal mucosal irritation, nausea, headache and vomiting.

The primary endpoint of the study was evidence of a chorionic sac in transvaginal sonography 21-23 days after IUI with a positive serum hCG test.

Statistical analysis was carried out using SPSS 16.0. Binary logistic regression was applied for calculation of Odds ratio and likelihood ratio test. For all comparisons, p < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for couples were idiopathic infertility, polycystic ovary syndrome (PCOS) and / or male subfertility.
* Age 18-42
* In all patients fallopian tubes were documented to be patent by sonographic contrast hysterosalpingography (Echovist® 200, Bayer Vital GmbH, Leverkusen, Germany) or by chromo-laparoscopy.
* Infections with Hepatitis B and C and HIV were excluded in all couples by negative serological tests.
* In all patients protective titers against rubella virus were confirmed.

Exclusion Criteria:

* Patients displaying signs or symptoms of anomalies such as uterine fusion defects, submucosal fibroids, active endometriosis or acute inflammation were excluded from the study.
* Further prerequisites were endocrine serum parameters (FSH, LH, estradiol, testosterone, SHBG, DHEA-S, Prolaktin, TSH) from cycle day 2-5 within the normogonadotropic range with no evidence of hyperandrogenemia, thyroid dysfunction or hyperprolactinemia. 1

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2003-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 1 month

SECONDARY OUTCOMES:
Possible side effects: nasal mucosal irritation, headake, lower abdominal pain | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Obstetrics and Gynecology, Munich, Germany